CLINICAL TRIAL: NCT03345706
Title: To Evaluate the Feasibility and Safety of Selective Cerebral Hypothermia in Out-of-hospital Cardiac Arrest (OHCA) Patients Receiving ECPR.
Brief Title: Selective Cerebral Hypothermia Trial - Under Extracorporeal Cardiopulmonary Resuscitation (SHOT-ECPR)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 201603049DIPA
Record Dates: First submitted 2017-10-30; First posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-10

CONDITIONS: Out-Of-Hospital Cardiac Arrest
Keywords: Hypothermia,ECPR
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Selective cerebral hypothermia (Experimental): Selective cerebral hypothermia
  Interventions: Procedure: Selective cerebral hypothermia
- Regular hypothermia (Active Comparator): Regular hypothermia
  Interventions: Procedure: Regular hypothermia

INTERVENTIONS:
Procedure: Selective cerebral hypothermia — Subjects will be transferred to ICU for the 12-hour selective cerebral hypothermia procedure. Cooling will be initiated and targeted to reach ipsilateral nasal temperature of 27±2°C for 12 hours, followed by controlled rewarming.
  Arms: Selective cerebral hypothermia
Procedure: Regular hypothermia — Subjects will be transferred to ICU for the 12-hour selective cerebral hypothermia procedure. Subjects will receive systemic hypothermia via ECMO at 33.5±0.5°C (33-34°C) for 48 hours at the same time.
  Arms: Regular hypothermia

SUMMARY:
The study is designed as a pilot, open-label study to investigate the feasibility and safety of selective cerebral hypothermia in OHCA patients receiving ECPR.

DETAILED DESCRIPTION:
Patients with OHCA and meeting the criteria for initiating extracorporeal membrane oxygenation (ECMO) criteria will be checked for eligibility for the study during CPR by the emergency physicians or staff at the scene. Informed consent will be asked as well. The standard V-A circuit for ECMO will be applied to the patients as soon as they arriving ER following the standard operation procedure of the hospital. The necessary testing and procedures will be applied to check the eligibility of the patients. Eligible subjects and/or their legal representatives will be further confirmed for the consent of experimental selective cerebral hypothermia. Systemic hypothermia at 33.5+/-0.5°C (33-34°C) for 48 hours will be performed to all eligible subjects.

For subjects who consent to receive selective cerebral hypothermia, they will be transferred to the catheterization lab for the blood flow controlling and cooling system settlement. Subjects then will be transferred to ICU for the 12-hour selective cerebral hypothermia procedure. Cooling will be initiated and targeted to reach ipsilateral nasal temperature of 27+/-2°C for 12 hours, followed by controlled rewarming. Both ipsilateral and contralateral nasal temperature will be monitored throughout. Activated clotting time (ACT) monitoring should be performed every 2 hours till stable and then every 12 hours during the whole cooling procedure. Also, subjects will receive systemic hypothermia via ECMO at 33.5+/-0.5°C (33-34°C) for 48 hours at the same time.

Subjects will stay and be observed in ICU until subject's condition is stable and can be transferred to general ward by investigator's judgment. The weaning of ECMO will be judged by investigator based on the subject's condition.

For subjects who do not agree to receive selective cerebral hypothermia, only the systemic hypothermia via ECMO will be applied. Subjects will receive systemic hypothermia at 33.5+/-0.5°C (33-34°C) for 48 hours via ECMO following the standard operative procedure.

Subject weaned from ECMO will be transferred to ward and will be followed until 6 months after the event. Outcome improvement and safety will be evaluated following scheduled timeline.

The study intends to enroll 20 subjects and is expected that 10 among the 20 enrolled subjects will receive selective cerebral hypothermia. The data from subjects who do not receive the experimental procedure will be used as the control group when data analyzing for the efficacy and safety of selective cerebral hypothermia.

ELIGIBILITY:
Main inclusion criteria:

Patients are eligible for inclusion in this study, if they fulfil all of the following criteria:

1. Clinical symptoms and signs compatible with OHCA.
2. Age between 20-65 years.
3. Eligible for initiating ECMO criteria.
4. No flow period less than 10 minutes.
5. CPR for longer than 10 minutes without return of spontaneous circulation (ROSC) under active CPR
6. Unconsciousness. Glasgow Coma Scale (GCS) 7T and M4 with tracheal tube 30 minutes after ECMO setup.
7. The ECMO flow can be maintained stable and return of spontaneous beating after ECMO setup for 2 hours.
8. The blood pressure can be maintained with mean pressure around 55 mmHg for 2 hours.
9. Patient or patient's legal representatives is willing to provide the signed informed consent.
10. Able to provide signed informed consent form (ICF) within 6 hours after the event and proceed to selective cerebral hypothermia within 12 hours after the event.

Main exclusion criteria:

Patients with any of the following characteristics must not be included in the study:

1. ROSC for 20 minutes after resuscitation without repeated collapse
2. Terminal stage malignancy
3. Pre-existing multi-organ dysfunction
4. Ventilator-dependent > 3 months
5. Bed-ridden > 3 months, not self-independent before CPR
6. Traumatic origin, uncontrollable bleeding
7. Patients with cerebral aneurysm
8. Patients with sepsis (blood culture positive)
9. Pregnancy
10. CT scan evidence of cerebral hemorrhage or non-ischemic etiology of neurologic symptoms
11. Severe, untreatable aortoiliac disease or small-caliber iliac arteries restricting vascular access with a 14 French sheath
12. Patients with either side common or internal carotid arteries >50% stenosis and cannot be worked around
13. Patient with "DNR" order

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-10-11 (Actual); Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
The feasibility and safety of selective cerebral hypothermia in out-of-hospital cardiac arrest (OHCA) patients receiving ECPR. | 12 hours
  The laboratory tests( CBC, liver function, kidney function, electrolytes,coagulation) . The percentage of subjects who have clinically-significant abnormal findings will be summarized by individual assessments of each category.

SECONDARY OUTCOMES:
The outcome of selective cerebral hypothermia in OHCA patients receiving ECPR. | 6 Month
  The laboratory tests (CBC, liver function, kidney function, electrolytes, coagulation) .The percentage of subjects who have clinically-significant abnormal findings will be summarized by individual assessments of each category.

CONTACTS AND LOCATIONS:
Overall Officials: Chen Yih-Sharng, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan